CLINICAL TRIAL: NCT04840264
Title: A Multi-center, Non-randomized, Three-cohort, Phase II Trial of a Modified Triplet Combination of Docetaxel, Oxaliplatin and Fluorouracil for Gastric Cancer With Peritoneal Carcinomatosis and Inoperable Malignant Bowel Obstruction
Brief Title: Docetaxel, Oxaliplatin and 5-FU for Gastric Cancer With Inoperable Malignant Bowel Obstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Doctor of Medicine, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhenJing
Record Dates: First submitted 2019-09-11; First posted 2021-04-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Peritoneal Carcinomatosis
Keywords: Malignant Bowel Obstruction; Docetaxel; Oxaliplatin; Fluorouracil
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Docetaxel; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (First-Line Therapy) (Experimental): Docetaxel 25 mg/square metre, ivdrip 60 min, D1, D8, D15; Oxaliplatin 85 mg/square metre, ivdrip 180 min, D1, D15; 5Fu 1200 mg/square metre, civ 24 hours, D1, D8, D15; Repeat every 4 weeks.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Fluorouracil
- B (Second-Line Therapy) (Experimental): Docetaxel 25 mg/square metre, ivdrip 60 min, D1, D8, D15; Oxaliplatin 85 mg/square metre, ivdrip 180 min, D1, D15; 5Fu 1200 mg/square metre, civ 24 hours, D1, D8, D15; Repeat every 4 weeks.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Fluorouracil
- C (Third- or Later-Line Therapy) (Experimental): Docetaxel 25 mg/square metre, ivdrip 60 min, D1, D8, D15; Oxaliplatin 85 mg/square metre, ivdrip 180 min, D1, D15; 5Fu 1200 mg/square metre, civ 24 hours, D1, D8, D15; Repeat every 4 weeks.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Docetaxel — 25 mg/square metre, D1, D8, D15, repeat every 4 weeks.
Drug: Oxaliplatin — 85 mg/msquare metre, D1, D15, repeat every 4 weeks.
Drug: Fluorouracil — 1200 mg/square metre, D1, D8, D15, repeat every 4 weeks.
  Other Names: 5-FU

SUMMARY:
This is a multi-center, non-randomized, 3-cohort, phase II trial, evaluating a triplet combination of docetaxel, oxaliplatin and fluorouracil for gastric cancer with peritoneal carcinomatosis and inoperable malignant bowel obstruction.

DETAILED DESCRIPTION:
The primary study hypothesis is that the regimen will provide a clinically meaningful bowel obstruction clearance. This trial has 3 paralleled cohorts with the same experimental regimen: Cohort A (first-line therapy) will include 35 participants who have not received any palliative chemotherapy; Cohort B (second-line therapy) will include 22 participants who progress after the first-line therapy; Cohort C (third- or later-line therapy) plans to include 22 cases who have received two or more prior therapies for their metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age;
* ECOG PS ≤3;
* pathologically diagnosed gastric or gastroesophageal junctional adenocarcinoma;
* peritoneal carcinomatosis established by imaging data or pathological evidence;
* MBO below the Treitz ligament based on clinical grounds or radiological findings;
* considered as inoperable MBO by two independent surgical consultants;
* Hb≥60g/L, WBC ≥4×10E9/L, ANC≥2×10E9/L，PLT≥100×10E9/L;
* Cr≤ Upper Normal Limit(UNL);
* Tbil≤1.5 UNL,AST≤1.5 UNL, ALT≤1.5 UNL, ALP≤1.5 UNL;
* Written informed consent form paticipants.

Exclusion Criteria:

* treated by a combination regimen containing all the study drugs;
* allergy to any of the study drugs;
* HER-2 amplification or overexpression, mismatch repair protein expression deletion (dMMR), or genetic testing suggestive of high microsatellite instability (MSI-H);
* strangulated intestinal obstruction;
* active gastrointestinal bleeding;
* uncontrolled active infection;
* unstable heart diseases with severe ECG abnormalities or affect clinical treatment (such as cardiac insufficiency, myocardial infarction, angina);
* severe lung diseases (such as interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc);
* mental disorders that affect clinical treatment or central nervous system diseases;
* concomitant cerebral parenchymal or meningeal metastasis;
* HIV infection or untreated active hepatitis;
* bowel surgery or stenting required due to obstruction;
* pregnant or lactating women;
* other conditions that are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
60-day Obstruction Clearance Rate | 60 days
  proportion of participants who achieved obstruction clearance within 60 days from start of treatment

SECONDARY OUTCOMES:
30-day Obstruction Clearance Rate | 30 days
  proportion of participants who achieved obstruction clearance within 30 days from start of treatment
Time to Obstruction Clearance | 60 days
  interval from start of treatment to obstruction clearance
Obstruction Clearance Duration | 2 years
  interval from obstruction clearance to the next malignant bowel obstruction
Safety in terms of Adverse Events | 2 years
  according to Common Terminology Criteria for Adverse Events version 5.0
Overall Survival | 2 years
  interval from start of treatment to death or last follow-up
Quality of Life assessed by EORTC QLQ-OG25 | 3 months
  in terms of European Organization for Research and Treatment of Cancer Quality of Life questionnair OG25

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, MD, Study Chair — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated hosipital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anthony T, Baron T, Mercadante S, Green S, Chi D, Cunningham J, Herbst A, Smart E, Krouse RS. Report of the clinical protocol committee: development of randomized trials for malignant bowel obstruction. J Pain Symptom Manage. 2007 Jul;34(1 Suppl):S49-59. doi: 10.1016/j.jpainsymman.2007.04.011. Epub 2007 Jun 4. PMID 17544243
- [Background] Madariaga A, Lau J, Ghoshal A, Dzierzanowski T, Larkin P, Sobocki J, Dickman A, Furness K, Fazelzad R, Crawford GB, Lheureux S. MASCC multidisciplinary evidence-based recommendations for the management of malignant bowel obstruction in advanced cancer. Support Care Cancer. 2022 Jun;30(6):4711-4728. doi: 10.1007/s00520-022-06889-8. Epub 2022 Mar 10. PMID 35274188